CLINICAL TRIAL: NCT06078410
Title: A Prospective Cohort Study of Neurologic Evaluation in Patients Recevied Transapical Beating-heart Septal Myectomy or General Cardiac Surgery
Brief Title: Neurologic Evaluation of Patients After Transapical Beating-Heart Septal Myectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiang Wei (Other)
Responsible Party: Sponsor-Investigator, Xiang Wei, Professor and Director, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2023-S034
Record Dates: First submitted 2023-09-27; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy (HOCM); Neurologic Evaluation; Magnetic Resonance Imaging (MRI); Transapical Beating-Heart Septal Myectomy; Cardiac Surgery Involving Left Heart Operation
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TA-BSM: patients received transapical beating-heart septal myectomy
  Interventions: Procedure: Cardiac surgery
- Cardiac surgery involving left heart operation: patients received cardiac surgery involving left heart operation, such as valvuloplasty, valve replacement, repair of auricular septal defect, repair of auricular/ventricular septal defect

INTERVENTIONS:
Procedure: Cardiac surgery — The TA-BSM group will undergo transapical beating-heart septal myectomy and the group of cardiac surgery involving left heart operation will udergo patients received cardiac surgery involving left heart operation, such as valvuloplasty, valve replacement, repair of auricular septal defect, repair of auricular/ventricular septal defect.
  Groups: TA-BSM

SUMMARY:
The goal of this prospective cohort study is to evaluate the neurologic changes in patients that received transapical beating-heart septal myectomy. The main questions are: whether this novel operation way would cause neurologic impairment; whether this novel operation way have similar neurologic lesions, compared to other cardiac surgery ways. Participants will undergo detailed neurologic and cognitive assessment at baseline, after procedure, and at 30 days. Researchers will compare the clinically relevant manifestations and brain lesions measured by cognitive evaluation forms of the nervous system (i.e. Montreal cognitive assessment) and diffusion-weighted magnetic resonance imaging (DW-MRI) to assess the safety of transapical beating-heart septal myectomy on nervous system.

DETAILED DESCRIPTION:
Nervous system complication is one of the common complications caused by cardiac surgery, including ischemic stroke, encephalopathy, neurocognitive dysfunction, which can increase the mortality of patients, hospitalization cost and lead to long-term quality of life impairment. At present, embolism is considered to be the main mechanism of postoperative nervous system complication. Imaging studies have confirmed that 30% to 50% of perioperative strokes are caused by brain embolism larger than 200 μm. For example, a study using diffusion-weighted magnetic resonance imaging (DW-MRI) found that 66% of patients who received aortic valve replacement had a new cerebral infarction with a brain injury volume of about 126 mm3. Recently, our team have invented a novel surgical method called transapical beating-heart septal myectomy (TA-BSM) to cure hypertrophic obstructive cardiomyopathy (HOCM). To date, this novel therapy displayed ideal effectiveness on these patients, however, whether this novel operation way would cause neurologic impairment is unclear. In this study, researchers will compare TA-BSM with cardiac surgery involving left heart operation, and analyze the clinically relevant manifestations and brain lesions measured by cognitive evaluation forms of the nervous system (i.e., Montreal cognitive assessment) and diffusion-weighted magnetic resonance imaging (DW-MRI) in these patients received above therapies. This study is to assess the safety of TA-BSM on nervous system and contributes the further improvement of this novel cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

meets indications for transapical beating-heart septal myectomy procedure or these cardiac surgery involving left heart operation, such as hypertrophic obstructive cardiomyopathy, mitral valve prolapse, and ventricular septal defect; willing to comply with protocol-specified follow-up evaluations.

Exclusion Criteria:

severe brain infarction, such stroke and cerebral hemorrhage recently; the implantation of metal materials, including Pacemaker; not able to undergo MRI examination; peptic ulcer or recent gastrointestinal bleeding (<6 months); the history of myocardial infarction; cognitive impairment in the past; not able to finish nervous system evaluation scale.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffer from hypertrophic obstructive cardiomyopathy or the other cardiovascular disease and have to receive cardiac surgery involving left heart operation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of diffusion-weighted MRI lesions | 3 months
  the number (n) of new brain lesions measured by diffusion-weighted magnetic resonance imaging (DW-MRI) in 3 months
The volume of new brain lesions measured by diffusion-weighted MRI | 3 months
  the volume (mL) of new brain lesions measured by diffusion-weighted magnetic resonance imaging (DW-MRI) in 3 months

SECONDARY OUTCOMES:
neurologic injury | 7 days and 3 months
  The number of participants (n) with neurological events and cognitive dysfunction following transapical beating-heart septal myectomy
all-cause and cardiovascular mortality | 7 days and 3 months
  all-cause and cardiovascular mortality following transapical beating-heart septal myectomy
montreal cognitive assessment | 7 days and 3 months
  montreal cognitive assessment evaluating mild cognitive impairment, ranging from 0 to 30, in which higher scores mean a better outcome.
national Institute of Health stroke scale | 7 days and 3 months
  national Institute of Health stroke scale evaluating mild cognitive impairment, ranging from 0 to 42, in which higher scores mean a worse outcome.
modified rankin scale | 7 days and 3 months
  modified rankin scale evaluating mild cognitive impairment, ranging from 0 to 6, in which higher scores mean a worse outcome.
symbol digit modalities test | 7 days and 3 months
  symbol digit modalities test evaluating mild cognitive impairmentt, ranging from 0 to 90, in which higher scores mean a better outcome.
trail-making-test | 7 days and 3 months
  trail-making-test evaluating mild cognitive impairment, in which the longer time mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Wei, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
All of the conclusive participant data, after removing the individual information of privacy, will be uploaded as supporting information when publishing the current study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the current study is published

REFERENCES:
- [Result] Fang J, Wang R, Liu H, Su Y, Chen J, Han X, Wei Y, Chen Y, Cheng L, Wei X. Transapical septal myectomy in the beating heart via a minimally invasive approach: a feasibility study in swine. Interact Cardiovasc Thorac Surg. 2020 Feb 1;30(2):303-311. doi: 10.1093/icvts/ivz249. PMID 31642911